CLINICAL TRIAL: NCT02904980
Title: A Randomised Controlled Trial of a Group-based, Gaze Training Intervention for Children With Developmental Coordination Disorder
Brief Title: The Effects of a Group-based Gaze Training Intervention for Children With Developmental Coordination Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manchester Metropolitan University (Other)
Collaborators: Liverpool Hope University (Other); University of Exeter (Other); University of Calgary (Other); The Waterloo Foundation (Other)
Responsible Party: Principal Investigator, Greg Wood, Lecturer in Sport and Exercise Psychology, Manchester Metropolitan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15/NW/0279
Record Dates: First submitted 2016-09-09; First posted 2016-09-19 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2016-09

CONDITIONS: Developmental Coordination Disorder
Keywords: Quiet eye training; Visual Attention
MeSH Terms: conditions — Motor Skills Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Technical Training Group (Experimental): 15 children diagnosed with DCD
  Interventions: Behavioral: Technical Training
- Quiet Eye Training Group (Experimental): 15 children diagnosed with DCD
  Interventions: Behavioral: Quiet Eye Training

INTERVENTIONS:
Behavioral: Technical Training — Children will watch an instructional video focused on movement related instructions regarding the throwing and catching task.
  Arms: Technical Training Group
Behavioral: Quiet Eye Training — Children will watch the same video as the TT group but will also receive instructions designed to optimise their quiet eye durations.
  Arms: Quiet Eye Training Group

SUMMARY:
The aim of this study was to integrate a gaze training intervention (i.e., quiet eye training; QET) that has been shown to improve the throwing and catching skill of children with Developmental Coordination Disorder (DCD), within an approach (i.e., group therapy) that might alleviate the psychosocial influence of these motor skill deficits.

DETAILED DESCRIPTION:
Children with DCD will be randomly split into either QET group or a technical training (TT). The TT group will be given movement-related instructions via video, relating to the throw and catch phases, while the QET group will also be taught to fixate a target location on the wall prior to the throw (QE1) and to track the ball prior to the catch (QE2). Each group will take part in a 4- week, group therapy intervention and measurements of QE duration obtained from a mobile eye tracking system and catching performance are to be taken before and after training, and at a 6-week delayed retention test. Parental feedback on psychosocial and motor skill outcomes will also be collected at delayed retention.

ELIGIBILITY:
Inclusion Criteria:

* Prior diagnosis of Developmental Coordination Disorder or suspected to have DCD
* Scores below the 5th percentile on the MABC-2 (Movement Assessment Battery for Children-2)
* Be of normal intelligence (assessed through parent/teacher feedback)
* No neurological disorder
* Normal of corrected-to-normal vision

Exclusion Criteria:

* Score over 5th Percentile on the MABC-2
* Suffers from a neurological disorder
* Below average intelligence
* Any visual impairment

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2015-02; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change in Catching Success | From Baseline to after a 4 week training period, and after 6-week delayed retention test
  How many balls the participants catch out of 50 attempts
Changes in the qualitative catching performance scale score | From Baseline to after a 4 week training period, and after 6-week delayed retention test
  The qualitative catching performance scale consisted of an 11-point scale whereby catch attempts were given a score between '0' (Makes no move towards the ball as it comes back) and '10' (The catch is made exclusively with the palms and fingers).
Changes in Quiet Eye durations | From Baseline to after a 4 week training period, and after 6-week delayed retention test
  Changes in participants eye-movements

SECONDARY OUTCOMES:
Changes 3D Movement Kinematics | From Baseline to after a 4 week training period, and after 6-week delayed retention test
  Changes in joint angles related to the throwing movement
Changes in Muscular Activity (EMG) | From Baseline to after a 4 week training period, and after 6-week delayed retention test
  Changes in muscular activity related to the throwing task
Parental Perceptions of Motor Skill Improvements | End of the study (approximately 12 weeks after baseline testing)
  Parent feedback will be gathered using a short answer questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Omid Alizadehkhaiyat, PhD, Study Director — Liverpool Hope University
Locations (1):
- Manchester Metropolitan University, Crewe, Cheshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miles CA, Wood G, Vine SJ, Vickers JN, Wilson MR. Quiet eye training facilitates visuomotor coordination in children with developmental coordination disorder. Res Dev Disabil. 2015 May;40:31-41. doi: 10.1016/j.ridd.2015.01.005. Epub 2015 Feb 25. PMID 25721344
- [Derived] Wood G, Miles CA, Coyles G, Alizadehkhaiyat O, Vine SJ, Vickers JN, Wilson MR. A randomized controlled trial of a group-based gaze training intervention for children with Developmental Coordination Disorder. PLoS One. 2017 Feb 10;12(2):e0171782. doi: 10.1371/journal.pone.0171782. eCollection 2017. PMID 28187138